CLINICAL TRIAL: NCT02879071
Title: Long Term Follow-up After Embolization of Brain Arteriovenous Malformations
Acronym: MAV-endovasc
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RBC_2015_17
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Arteriovenous Malformations
MeSH Terms: conditions — Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
The time-frame and the follow-up elements after embolization of brain arteriovenous malformations are not standardized. Therefore, few reliable follow-up data are available for these patients. This study aims at collecting standardized long term data for these patients.

ELIGIBILITY:
Inclusion Criteria:

* arteriovenous malformation
* age > 18 years old

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing embolization for an arteriovenous malformation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-11-26 (Actual); Primary Completion 2037-11-25 (Estimated); Study Completion 2037-11-25 (Estimated)

PRIMARY OUTCOMES:
angiographic evaluation of the arteriovenous malformation occlusion | 5 years after embolization

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] Baharvahdat H, Blanc R, Fahed R, Pooyan A, Mowla A, Escalard S, Delvoye F, Desilles JP, Redjem H, Ciccio G, Smajda S, Hamdani M, Mazighi M, Piotin M. Endovascular treatment as the main approach for Spetzler-Martin grade III brain arteriovenous malformations. J Neurointerv Surg. 2021 Mar;13(3):241-246. doi: 10.1136/neurintsurg-2020-016450. Epub 2020 Sep 28. PMID 32989031
- [Derived] Baharvahdat H, Blanc R, Fahed R, Smajda S, Ciccio G, Desilles JP, Redjem H, Escalard S, Mazighi M, Chauvet D, Robert T, Sasannejad P, Piotin M. Endovascular Treatment for Low-Grade (Spetzler-Martin I-II) Brain Arteriovenous Malformations. AJNR Am J Neuroradiol. 2019 Apr;40(4):668-672. doi: 10.3174/ajnr.A5988. Epub 2019 Feb 21. PMID 30792251